CLINICAL TRIAL: NCT01500538
Title: A Pilot Study of Oral Vorinostat Plus Oral Eltrombopag Support in Patients With Lymphoma (VEIL)
Acronym: VEIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment rate
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/111
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2012-10

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma
Keywords: Follicular lymphoma; Marginal zone lymphoma; Mantle cell lymphoma; thrombocytopenia; eltrombopag; vorinostat; lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Thrombocytopenia; Lymphoma | interventions — eltrombopag; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag and vorinostat combination therapy (Experimental): Daily oral intake of 400mg vorinostat if necessary with combination therapy eltrombopag commencing at 50mg per day increasing to a maximum of 200mg per day
  Interventions: Drug: Eltrombopag and Vorinostat

INTERVENTIONS:
Drug: Eltrombopag and Vorinostat — 4 week mono-therapy eltrombopag, commencing at 50mg/day, increasing to 200mg. Daily intake of 400mg vorinostat for minimum of 6 cycles, each cycle of 4 weeks, possibly in combination with daily intake eltrombopag commencing at 50mg/day at a maximum dose of 200md/day (150mg/day for subjects of East-Asian ancestry)
  Other Names: Revolade (eltrombopag); Zolinza (vorinostat)

SUMMARY:
Vorinostat is a drug (Histone Deacetylase Inhibitor [HDACi]) administered orally that has been approved in United States for the patients with cutaneous Tcell lymphoma (CTCL) who have progressive, persistent or recurrent disease on or following two systemic therapies.

In the early period of treatment with vorinostat, some patients may experience low platelet counts. Therefore this study will be examining the combination of these two medications (Vorinostat and eltrombopag) to assess if eltrombopag can overcome the low platelets during treatment with vorinostat.

Eltrombopag is a drug administered orally designed to mimic the protein thrombopoietin, which causes the body to make more platelets. Eltrombopag has been registered in Australia and approved overseas to treat patients with chronic ITP (Immune Thrombocytopenia Purpura) a disease where patients destroy their own platelets very rapidly and thus develop low platelet count) but it is not registered and it is not yet known whether eltrombopag can increase platelet counts in patients treated with the HDACi.

The aim of this project is to test whether Vorinostat and eltrombopag can be safely combined, and to test whether they are effective in participants with T-cell lymphoma involving the skin or patients with relapsed/refractory follicular lymphoma (FL), marginal zone lymphoma (MZL), or mantle cell lymphoma (MCL)

A total of 25 people with Cutaneous T cell lymphoma/ CTCL, marginal zone lymphoma, follicular lymphoma or mantle cell lymphoma will be recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18years or older
* T-cell lymphoma involving the skin or patients with relapsed/refractory follicular lymphoma (FL), marginal zone lymphoma (MZL), or mantle cell lymphoma (MCL). Disease must have been confirmed by previous histology and must be measurable
* For patients with cutaneous T-cell lymphoma: At least 2 prior systemic therapies (including 1 month of therapy with systemic steroids >25mg alternating days of prednisolone or equivalent, or total skin electron-beam radiotherapy). For patients with B cell lymphoma, prior exposure to a chemotherapy regimen is required, unless the patient is deemed to be unfit for conventional chemo-therapeutic regimens.
* Adequate haematological function: ANC ≥ 1.0x109/L
* Adequate renal function (serum creatinine clearance calculated as CrCl ≥30mL/min (perform 24hr urine creatinine clearance if serum creatinine is >1.5xULN);electrolyte levels ≥ LLN (i.e.: potassium, total calcium [corrected for serum albumin], magnesium and phosphorus) or correctable with supplements)
* Adequate hepatic function:AST and ALT ≤ 2.5 x ULN (or ≤ 5.0 x ULN if liver infiltration;Serum bilirubin ≤ 1.5 x ULN
* Life expectancy ≥ 12 weeks
* Written informed consent obtained prior to any study specific screening procedures
* ECOG performance status grade 0-2
* Ability to comply with adequate contraception in patients of childbearing potential.
* Females of childbearing potential must have had a negative urine pregnancy test at screening and agree to use a medically reliable method of preventing conception throughout the study and for 30 days following the date of last dose.
* Males with a female partner of childbearing potential must agree to use a medically reliable method of preventing conception throughout the study and for 30 days following the date of last dose.
* Mentally competent and is able to understand the information given and provide informed consent.

Exclusion Criteria:

* Known uncontrolled medical conditions which may compromise participation in this study including but not limited to:Poorly controlled congestive heart failure: ejection fraction <30% measured in past 6 months) or NYHA class IV;Unstable angina or an ischaemic cardiac event requiring hospital admission in the previous 12 months.
* Concomitant use of another HDAC inhibitor, including sodium valproate.
* GI disease that may significantly alter the absorption of eltrombopag
* Subjects known to be seropositive for HIV, Hepatitis B or Hepatitis C.
* Current participation in other trials or studies of medical therapeutic interventions.
* Known pro-thrombotic condition as defined by a history ≥1 unprovoked deep venous thrombosis or pulmonary embolism, or any DVT/PE with a procoagulant condition screen suggesting the presence of a procoagulant condition (prothrombin gene mutation homozygosity, factor V Leiden homozygosity, antithrombin deficiency, lupus anticoagulant syndrome).
* History of ischaemic neurological event (TIA or stroke) within the preceding 2 years.
* Active or uncontrolled infection, other than cutaneous infection.
* Prior diagnosis of cancer that was:more than 5 years prior to current diagnosis with subsequent evidence of disease recurrence or estimated clinical expectation of recurrence is greater than 10% within next 2 years;within 5 years of current diagnosis with the exception of successfully treated basal cell or squamous cell skin carcinoma, carcinoma in situ of the cervix or localised cancer treated curatively with local therapy only
* Use of another anti-cancer treatment within 21 days of starting vorinostat, with the exception of steroids, interferon or oral methotrexate which have been at a stable dose for at least 4 weeks prior to day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The occurrence of all grade III/IV adverse events (haematological and non haematological) during vorinostat and eltrombopag combination therapy | One year from trial entry
  The period of observation for the primary endpoint is defined as the observation for 6 cycles of eligible patients who have commencement eltrombopag following commencement of vorinostat.

SECONDARY OUTCOMES:
Occurrence of thrombocytopenia (TCP) with vorinostat therapy and response to eltrombopag: platelet, transfusion and bleeding endpoints | One year from trial entry
  Occurrence & severity of thrombocytopenia (TCP), all grades at baseline & during first 6 vorinostat cycles.
  Occurrence & severity of worsening grade of TCP (relative to day 1 cycle 1 of vorinostat therapy) after cycle 1 day 8.
  Occurrence & severity of TCP following withdrawal of eltrombopag in patients who had protocol-specified withdrawal of eltrombopag.
  Occurrence of platelet response, defined as a cycle nadir platelet count showing a 50% improvement in platelet nadir compared to previous cycle & at least an absolute increase of 20x109/L.
  Occurrence of grade III/IV TCP during vorinostat treatment cycle among patients who experience a platelet nadir ≤25 x109/L, receive eltrombopag & who then achieve a platelet response.
  Percentage drop in platelet count from day 1 of cycle to nadir & percentage drop in neutrophil count from day 1 of cycle to nadir, for each cycle.
  Occurrence & severity of clinically significant bleeding events defined as per the WHO bleeding scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, MBBS (Hons), FRCPA, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia